CLINICAL TRIAL: NCT04084678
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study of Ralinepag to Evaluate Safety and Effects on Exercise Capacity Assessed by CPET in Subjects With WHO Group 1 Pulmonary Hypertension Who Recently Initiated Therapy
Brief Title: A Study of Ralinepag to Evaluate Effects on Exercise Capacity by CPET in Subjects With WHO Group 1 PH
Acronym: CAPACITY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROR-PH-302
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: PAH; Pulmonary Hypertension; Hypertension; Connective Tissue Disease; Familial Primary Pulmonary Hypertension; Vascular Diseases; Cardiovascular Diseases; Hypertension, Pulmonary; Lung Diseases; Respiratory Tract Disease; Pulmonary Arterial Hypertension
Keywords: Prostacyclin; Connective Tissue Disease-Associated; Cardiopulmonary Exercise Capacity (CPET); IP Receptor Agonist
MeSH Terms: conditions — Hypertension, Pulmonary; Hypertension; Connective Tissue Diseases; Familial Primary Pulmonary Hypertension; Vascular Diseases; Cardiovascular Diseases; Lung Diseases; Respiratory Tract Diseases; Pulmonary Arterial Hypertension | interventions — ralinepag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ralinepag (Experimental): Ralinepag once daily extended-release tablets (oral) 50, 250, and 400 mcg titrated to the individual maximum tolerated dose (maximum dose of 1400 mcg)
  Interventions: Drug: Ralinepag
- Placebo (Placebo Comparator): Matching placebo tablets (oral)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ralinepag — Oral ralinepag
  Other Names: APD811
  Arms: Ralinepag
Drug: Placebo — Matching oral tablets
  Arms: Placebo

SUMMARY:
Study ROR-PH-302, ADVANCE CAPACITY, is designed to evaluate the effects of ralinepag therapy on exercise capacity as assessed by change in peak oxygen consumption (VO2) derived from cardiopulmonary exercise testing (CPET) after 28 weeks of treatment

DETAILED DESCRIPTION:
ROR-PH-302 is a 28-week multicenter, randomized, double-blind, placebo-controlled study. Subjects who meet entry criteria will be randomly allocated 2:1 to receive ralinepag or placebo, in addition to their PAH-specific background therapy, as applicable. The primary endpoint is change from Baseline in peak VO2 (assessed by CPET) at Week 28. All subjects who complete the study on study drug through Week 28 will have the option to receive ralinepag in an open-label extension (OLE) study. Subjects who discontinue study drug prior to Week 28, as well as those who complete Week 28 on study drug but choose not to participate in the OLE study, will be contacted every 6 months and at the end of the study to determine their survival status. Subjects who prematurely discontinue study drug or withdraw from the study for any reason will not be eligible to enter the OLE study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. At least 18 years of age.
3. Primary diagnosis of PAH.
4. Has had a diagnostic RHC performed at or within 3 years before Screening (or at Screening if one is not available) that is consistent with the diagnosis of PAH.
5. Has World Health Organization (WHO)/New York Heart Association (NYHA) Functional Class (FC) II to III symptoms
6. Must be on a stable dose of PAH-specific oral therapy, defined as no change in dose or regimen for at least 90 days prior to randomization. Allowable PAH-specific therapy is an endothelin receptor antagonist and/or a phosphodiesterase type 5 inhibitor (PDE5-I) or a soluble guanylate cyclase (sGC) stimulator. Subjects may be on a stable dose of either a PDE5-I or a sGC stimulator, not both.
7. Has a 6-minute walk distance (6MWD) of ≥150 meters at Screening.
8. Has a peak VO2 of ≥9 to <18 mL/min/kg during the Screening CPET, as assessed by the CPET core laboratory.
9. If the subject is taking concomitant medications that may affect the clinical manifestations of PAH, the subject must be on a stable dose for at least 30 days prior to randomization. The exception is that the dose of diuretics must be stable for at least the 10 days prior to randomization.
10. Both male and female subjects agree to use a highly effective method of birth control throughout the entire study period from informed consent through to the Week 28 Visit/28-day Follow-up Visit, if the possibility of conception exists. Eligible male and female subjects must also agree not to participate in a conception process during the study and for 30 days after the final dose of study drug. Eligible male subjects must agree not to participate in sperm donation for 90 days after the final dose of study drug. Women who are surgically sterile or postmenopausal are not considered to be of childbearing potential. If of childbearing potential, female partners of male study participants should agree to utilize medically acceptable methods of contraception for the duration of study participation.

Exclusion Criteria:

1. For subjects with known human immunodeficiency virus-associated PAH, a cluster of differentiation 4 T-cell count <200/mm3 at Screening.
2. Has 3 or more left ventricular disease/dysfunction risk factors.
3. Symptomatic coronary artery disease and/or myocardial infarction within past 6 months.
4. Current symptomatic aortic or mitral valve disease.
5. Has evidence of more than mild lung disease on pulmonary function tests performed within 1 year prior to, or during, Screening.
6. Has evidence of thromboembolic disease as determined by ventilation-perfusion lung scan or local standard of care diagnostic evaluation at or after diagnosis of PAH.
7. Current diagnosis of ongoing and clinically significant sleep apnea as defined by the Investigator.
8. Requires use of supplemental oxygen during CPET.
9. Respiratory exchange ratio <1.0 at Screening CPET as determined by the CPET core laboratory.
10. Acute non-cardiac disorder that may affect exercise performance or be aggravated by exercise (eg, infection, renal failure, thyrotoxicosis).
11. Male subjects with a QTcF >450 msec and female subjects with a QTcF >470 msec on electrocardiogram (ECG) recorded at Screening and analyzed by the central ECG laboratory. Subjects with evidence of intraventricular conduction delay, defined as a QRS interval >110 msec, will be excluded if QTcF is >500 msec for both males and females.
12. Severe chronic liver disease (ie, Child-Pugh Class C), portal hypertension, cirrhosis, or complications of cirrhosis/portal hypertension (eg, history of variceal hemorrhage, encephalopathy).
13. Confirmed active infection with hepatitis B virus or hepatitis C virus.
14. Subjects with alanine aminotransferase or aspartate aminotransferase ≥3 times the upper limit of normal or total bilirubin ≥2 times the upper limit of normal at Screening.
15. Chronic renal insufficiency as defined by an estimated glomerular filtration rate using the Modification of Diet in Renal Disease Study equation of <30 mL/min/1.73 m2 or requiring dialysis at Screening.
16. Hemoglobin concentration <9 g/dL at Screening.
17. Subjects treated with an intravenous, subcutaneous, inhaled, or oral prostacyclin pathway agent (eg, epoprostenol, treprostinil, iloprost, beraprost, or selexipag) for PAH within 90 days of randomization (use in vasoreactive testing is permitted). Subject is not eligible if previous prostacyclin therapy was stopped for a safety or tolerability issue related to systemic prostacyclin adverse effects.
18. Subject has pulmonary veno-occlusive disease.
19. Malignancy diagnosed and/or treated within 3 years of Screening, with the exception of localized non-metastatic basal cell or squamous cell carcinoma of the skin or in-situ carcinoma of the cervix excised with curative intent.
20. Subject tests positive for amphetamine, cocaine, methamphetamine, methylenedioxymethamphetamine, or phencyclidine in urine drug screen performed at Screening, or has a recent history (6 months) of alcohol or drug abuse. Subjects will not be excluded due to a positive drug screen caused by prescribed medications.
21. Initiation or discontinuation of a cardio-pulmonary rehabilitation program based upon exercise within 90 days prior to Screening and/or planned during study participation.
22. Prior participation in any study of ralinepag or another interventional clinical study with medicinal products within 30 days prior to Screening. Concurrent participation in registry or observational studies is allowed, if the subject can fulfill all other entry criteria and comply with all study procedures.
23. Any reason that, in the opinion of the Investigator, precludes the subject from participating in the study (eg, any previous or intercurrent medical condition) that may increase the risk associated with study participation or that would confound study analysis (eg, right-to-left shunt detected during CPET) or impair study participation or cooperation.
24. Known hypersensitivity to ralinepag or any of the excipients.
25. Life expectancy <12 months based on the Investigator's opinion.
26. Women who are pregnant, lactating, or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in peak VO2 assessed by CPET | Baseline to Week 28
  Peak VO2 by CPET was measured at Baseline (prior to starting study drug) and Week 28

SECONDARY OUTCOMES:
Change from Baseline in N-terminal pro-brain natriuretic peptide (NT-proBNP) | Baseline to Week 28
  NT-proBNP was measured at Baseline (prior to starting study drug) and Weeks 4, 8, 12, 16, 20, 24 and 28
Change from Baseline in Minute Ventilation (VE)/Carbon Dioxide output (VCO2) slope | Baseline to Week 28
  VE/VCO2 slope (from CPET) was calculated at Baseline (prior to starting study drug) and Week 28
Change from Baseline in health-related quality of life measured by the Short Form Health Survey (SF-36) Scores | Baseline to Week 28
  SF-36 was assessed at Baseline (prior to starting study drug) and Weeks 16 and 28. The SF-36 consisted of 36 questions in 8 health categories (Vitality, Physical Functioning, Bodily Pain, General Health Perception, Role Physical, Role Emotional, Social Functioning, and Mental Health). Responses to the questions were graded on a numerical scale, with 1 as the best score and higher numbers as worse scores. The raw scores from the subscales were converted and summed by the Investigator to a total score between 0 and 100 to measure functional health and well-being from the patient's point of view. The final score range was 0 (representing the lowest possible score; worst health state) to 100 (representing the highest possible score; best health state).
Time to First All-cause Non-elective Hospitalization | Baseline to Week 28
  The time to first all-cause nonelective hospitalization during the study period will be assessed.

CONTACTS AND LOCATIONS:
Locations (33):
- United States (5):
  - Banner University Medical Center (University of Arizona), Tucson, Arizona
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Tampa General Hospital/University of South Florida Center for Advanced Lung Disease and Lung Transplant, Tampa, Florida
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
- Argentina (2):
  - Hospital Britanico de Buenos Aires, Ciudad Autónoma de Bs. As.
  - Instituto de Cardiología de Corrientes, Corrientes
- Australia (4):
  - Macquarie University, North Ryde, New South Wales
  - Westmead Hospital, Dept Respiratory and Sleep Medicine, Westmead, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
- Austria (2):
  - Ordensklinikum Linz GmbH, Elisabethinen, Linz
  - AKH Wien, Innere Med. II, Kardiologie, Vienna
- Belgium (2):
  - Erasme University Hospital - Department of Cardiology, Brussels
  - Gasthuisberg University Hospital - Department of Pulmonology, Leuven
- Brazil (4):
  - Hospital Madre Teresa, Belo Horizonte, Minas Gerais
  - Hospital Sao Paulo, São Paulo, São Paulo
  - Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina de São Paulo - InCor-HCFMUSP, São Paulo, São Paulo
  - Centro de Hipertensão Pulmonar, Porto Alegre
- Canada (3):
  - Peter Lougheed Center, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - London Health Science Centre- Victoria Hospital, London, Ontario
- Germany (2):
  - Thoraxklinik-Heidelberg, Zentrum für Pulmonale Hypertonie, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Carl Gustav Carus TU Dresden, Medizinische Klinik I, Abteilung für Pneumologie, Dresden, Saxony
- Italy (3):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Centro Cardiologico Monzino, IRCCS, Milan
  - AOU Policlinico Umberto I, Rome
- Poland (2):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Klinika Kardiologii z Oddziałem Intensywnego Nadzoru Kardiologicznego, Bialystok
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina, Oddział Kardiologiczny, Otwock
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic I Provincial de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Imperial college Healthcare NHS Trust, London, United Kingdom